CLINICAL TRIAL: NCT02545075
Title: A Randomized, Open-Label, Two-arm, Comparative Study in Chinese Subjects With Chemotherapy Naïve Stage IV Melanoma Receiving Ipilimumab (3 mg/kg) vs. Dacarbazine
Brief Title: A Comparative Study in Chinese Subjects With Chemotherapy Naïve Stage IV Melanoma Receiving Ipilimumab (3 mg/kg) vs. Dacarbazine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-248
Record Dates: First submitted 2015-08-25; First posted 2015-09-09 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ipilimumab (Experimental): Intravenously (IV) 3 mg/kg every 3 weeks (at week 1,4,7,10) and thereafter (q3w/4 doses) at the time of progression
  Interventions: Drug: Ipilimumab
- Dacarbazine (Experimental): IV solution 250 mg/m2 (Day 1-5, every 3weeks/at week 1, 4, 7, 10,13,16,19,22)
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Ipilimumab
  Other Names: MDX-010
  Arms: Ipilimumab
Drug: Dacarbazine
  Other Names: DTIC
  Arms: Dacarbazine

SUMMARY:
The purpose of this study is to determine whether Ipilimumab will extend the life of chinese patients with Chemotherapy Naive Stage IV Melanoma more than Dacarbazine as well as to examine safety in this patient population.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Chinese males and females ≥ 18 years of age
* Histologic diagnosis of malignant melanoma
* Chemotherapy naive Stage IV melanoma (AJCC 2010)
* Life expectancy of ≥ 16 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Evidence of brain metastases on brain imaging
* Primary ocular or mucosal melanoma
* Any other malignancy from which the patient has been disease-free for less than 5 years
* BRAF status cannot be determined by Screening test
* Human Immunodeficiency Virus (HIV) positive or hepatitis B surface antigen (HBsAg) positive, or active Hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2015-10-31 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- China (8):
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Xi’an, Shanxi
  - Local Institution, Tianjin, Tianjin Municipality
  - Local Institution, Hanghzou, Zhejiang
  - Local Institution, Beijing
  - Local Institution, Kunming
  - Local Institution, Shanghai

REFERENCES:
- See also: BMS clinical trial educational resource — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 182 participants were enrolled, 68 were not randomized, reasons for not being randomized:3 participants withdrew consent and 65 no longer meet study criteria.
Groups:
- Ipilimumab (3 mg/kg): Ipilimumab 3 mg/kg to be administered via intravenous infusion over 90 minutes at Weeks 1, 4, 7 and 10, for a total of four doses in Induction (and Re-Induction for those randomized to the ipilimumab arm who qualify)
- Dacarbazine (250 mg/m2): DTIC 250 mg/m2 - Day 1 - 5, to be administered via intravenous infusion at Weeks 1, 4, 7, 10, 13, 16,19, and 22.
Period: Randomization
Arm/Group | Ipilimumab (3 mg/kg) | Dacarbazine (250 mg/m2)
Started (Partipants who were randomized) | 122 | 60
Completed (participants who were treated) | 122 | 53
Not Completed | 0 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 6
Period: Treatment
Arm/Group | Ipilimumab (3 mg/kg) | Dacarbazine (250 mg/m2)
Started (Participants who were treated) | 122 | 53
Completed (Participants who were continuing treatment period) | 0 | 0
Not Completed | 122 | 53
Not completed — Disease progression | 71 | 32
Not completed — Participant dicontinued study treatment | 7 | 9
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse event not related to study drug | 1 | 0
Not completed — Death | 1 | 0
Not completed — Participant drug toxicity | 1 | 0
Not completed — Completed treatment | 40 | 12

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab (3 mg/kg) | Dacarbazine (250 mg/m2) | Total
Number analyzed (Participants) | 122 | 60 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All randomized participants
  years | 53.6 (13.69) | 54.3 (13.39) | 53.8 (13.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 26 | 79
  Male | 69 | 34 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 122 | 60 | 182
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 122 | 60 | 182
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Two-Years Survival Rate
Description: Two-year survival rate is defined as the probability that a subject is alive at 2 years following the randomization date and will be estimated via the Kaplan-Meier (KM) method.
Time Frame: 24 months
Population: All randomized participants
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ipilimumab (3 mg/kg) | Dacarbazine (250 mg/m2)
Number analyzed (Participants) | 122 | 60
Percentage of Participants | 33.98 [28.36 to 39.67] | 34.09 [25.72 to 42.62]
Statistical Analysis 1: Comparison: Ipilimumab (3 mg/kg) vs Dacarbazine (250 mg/m2); Test type: Superiority; p = 0.5059, Chi-squared; One-sided p-value based on unstratified chi-square test

2. Secondary Outcome: One-Year Survival Rate
Description: Survival rate at 1 year is defined as the probability that a subject is alive at 1 year following the randomization date and will be estimated via the Kaplan-Meier (KM) method.
Time Frame: Approximately 43 months
Population: All randomized participants
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ipilimumab (3 mg/kg) | Dacarbazine (250 mg/m2)
Number analyzed (Participants) | 122 | 60
Percentage of Participants | 61.68 [55.71 to 67.09] | 64.11 [54.99 to 71.87]
Statistical Analysis 1: Comparison: Ipilimumab (3 mg/kg) vs Dacarbazine (250 mg/m2); Test type: Superiority; p = 0.6202, Chi-squared; One-sided unstratified chi-square

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined for each subject as the time between randomization date and the date of death (of any cause).
Time Frame: Approximately 43 months
Population: All randomized participants
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Ipilimumab (3 mg/kg) | Dacarbazine (250 mg/m2)
Number analyzed (Participants) | 122 | 60
Months | 15.08 [12.91 to 16.10] | 14.55 [13.37 to 19.19]
Statistical Analysis 1: Comparison: Ipilimumab (3 mg/kg) vs Dacarbazine (250 mg/m2); Test type: Superiority; p = 0.7267, Log Rank; One-sided p-value from Log-rank Test stratified by M substage (M1a+M1b vs. M1c); Stratified cox proportional hazard model = 1.13, 80% CI 2-sided [0.87 to 1.45]

4. Secondary Outcome: Progression Free Survival ( PFS)
Description: PFS is defined for each subject as the time between randomization date and the date of progression or death, whichever occurs first.
Time Frame: Approximately 43 months
Population: All randomized participants
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Ipilimumab (3 mg/kg) | Dacarbazine (250 mg/m2)
Number analyzed (Participants) | 122 | 60
Months | 2.60 [2.60 to 2.63] | 1.84 [1.41 to 2.63]
Statistical Analysis 1: Comparison: Ipilimumab (3 mg/kg) vs Dacarbazine (250 mg/m2); Test type: Superiority; p = 0.2503, Log Rank; One-sided p-value from Log-rank Test stratified by M substage (M1a+M1b vs. M1c) and BRAF mutation status as entered into the IVRS; Stratified Cox proportional hazard = 0.90, 80% CI 2-sided [0.71 to 1.15]

5. Secondary Outcome: Disease Control Rate ( DCR )
Description: Primary DCR is defined as the number of subjects in the arm with Best Overall Response (BOR) of complete response (CR), partial response (PR), or stable disease (SD), divided by the total number of randomized subjects in the arm.
Time Frame: Approximately 43 months
Population: All randomized participants
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab (3 mg/kg) | Dacarbazine (250 mg/m2)
Number analyzed (Participants) | 122 | 60
Percentage of participants | 32 [26.4 to 38.0] | 31.7 [23.7 to 40.6]
Statistical Analysis 1: Comparison: Ipilimumab (3 mg/kg) vs Dacarbazine (250 mg/m2); Test type: Superiority; p = 0.9932, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.00, 80% CI 2-sided [0.64 to 1.55]

6. Secondary Outcome: Best Overall Response Rate ( BORR )
Description: BORR definition is defined as the number of subjects in the arm with a BOR of CR or PR, divided by the total number of randomized subjects in the arm.
Time Frame: Approximately 43 months
Population: All randomized participants
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab (3 mg/kg) | Dacarbazine (250 mg/m2)
Number analyzed (Participants) | 122 | 60
Percentage of participants | 8.2 [5.2 to 12.3] | 8.3 [4.1 to 14.9]
Statistical Analysis 1: Comparison: Ipilimumab (3 mg/kg) vs Dacarbazine (250 mg/m2); Test type: Superiority; p = 0.9738, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.98, 80% CI 2-sided [0.48 to 2.03]

7. Secondary Outcome: Duration of Response ( DoR)
Description: DoR definition for the response evaluable subjects whose BOR is CR or PR is defined as the time between the date of response of CR or PR (whichever occurs first) and the first date of progressive disease (PD) or the date of death (whichever occurs first).
Time Frame: Approximately 43 months
Population: All randomized participants with response
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Ipilimumab (3 mg/kg) | Dacarbazine (250 mg/m2)
Number analyzed (Participants) | 10 | 5
Months | 8.99 [4.76 to 29.01] | 7.98 [1.45 to NA] — Upper limit had not be reached

8. Secondary Outcome: Duration of Stable Disease ( DoSD )
Description: Primary duration of stable disease (DoSD) definition for the randomized subjects whose BOR is SD is defined as the time between the randomization date and the first date of PD or the date of death (whichever occurs first)."
Time Frame: Approximately 43 months
Population: All randomized participants with BOR as stable disease
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Ipilimumab (3 mg/kg) | Dacarbazine (250 mg/m2)
Number analyzed (Participants) | 29 | 14
Months | 6.83 [5.29 to 7.62] | 9.40 [5.26 to 16.30]

ADVERSE EVENTS:
Time Frame: Approximately 43 months
Description: Adverse events are reported between first dose and 90 days after last dose of study therapy.
Groups:
- Ipilimumab: Ipilimumab 3 mg/kg to be administered via intravenous infusion over 90 minutes at Weeks 1, 4, 7 and 10, for a total of four doses in Induction (and Re-Induction for those randomized to the ipilimumab arm who qualify)
- Dacarbazine: DTIC 250 mg/m2 - Day 1 - 5, to be administered via intravenous infusion at Weeks 1, 4, 7, 10, 13, 16,19, and 22.
Arm/Group | Ipilimumab | Dacarbazine
All-Cause Mortality (participants affected / at risk) | 93/122 | 39/53
Serious Adverse Events (participants affected / at risk) | 34/122 | 12/53
Other Adverse Events (participants affected / at risk) | 118/122 | 48/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=122) | Dacarbazine (N=53)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 | 7
Cerebral infarction (Nervous system disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=122) | Dacarbazine (N=53)
Anaemia (Blood and lymphatic system disorders) | 8 | 3
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Sinus bradycardia (Cardiac disorders) | 4 | 3
Supraventricular tachycardia (Cardiac disorders) | 8 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 4
Constipation (Gastrointestinal disorders) | 14 | 14
Diarrhoea (Gastrointestinal disorders) | 7 | 4
Gastrointestinal disorder (Gastrointestinal disorders) | 4 | 8
Nausea (Gastrointestinal disorders) | 18 | 22
Vomiting (Gastrointestinal disorders) | 14 | 5
Asthenia (General disorders) | 12 | 8
Fatigue (General disorders) | 11 | 6
Oedema peripheral (General disorders) | 7 | 2
Pain (General disorders) | 15 | 6
Pyrexia (General disorders) | 23 | 10
Liver injury (Hepatobiliary disorders) | 1 | 5
Alanine aminotransferase increased (Investigations) | 31 | 19
Aspartate aminotransferase increased (Investigations) | 22 | 17
Bilirubin conjugated increased (Investigations) | 9 | 5
Blood albumin decreased (Investigations) | 15 | 5
Blood alkaline phosphatase increased (Investigations) | 6 | 4
Blood bilirubin increased (Investigations) | 14 | 5
Blood bilirubin unconjugated increased (Investigations) | 7 | 1
Blood chloride decreased (Investigations) | 7 | 5
Blood cholesterol increased (Investigations) | 6 | 4
Blood glucose increased (Investigations) | 10 | 5
Blood lactate dehydrogenase increased (Investigations) | 28 | 3
Blood potassium decreased (Investigations) | 1 | 3
Blood sodium decreased (Investigations) | 9 | 6
Blood thyroid stimulating hormone decreased (Investigations) | 11 | 0
Blood thyroid stimulating hormone increased (Investigations) | 27 | 4
Blood triglycerides increased (Investigations) | 15 | 5
Blood uric acid increased (Investigations) | 7 | 3
Blood urine present (Investigations) | 2 | 3
C-reactive protein increased (Investigations) | 25 | 4
Electrocardiogram T wave abnormal (Investigations) | 8 | 3
Gamma-glutamyltransferase increased (Investigations) | 17 | 11
Haemoglobin decreased (Investigations) | 22 | 6
Lymphocyte count decreased (Investigations) | 2 | 3
Neutrophil count decreased (Investigations) | 6 | 8
Neutrophil count increased (Investigations) | 16 | 2
Neutrophil percentage decreased (Investigations) | 7 | 1
Neutrophil percentage increased (Investigations) | 11 | 0
Platelet count decreased (Investigations) | 3 | 5
Platelet count increased (Investigations) | 13 | 1
Protein urine present (Investigations) | 4 | 4
Thyroxine free decreased (Investigations) | 7 | 1
Thyroxine free increased (Investigations) | 8 | 0
Tri-iodothyronine decreased (Investigations) | 7 | 0
Tri-iodothyronine free decreased (Investigations) | 9 | 0
Tri-iodothyronine free increased (Investigations) | 7 | 0
Weight decreased (Investigations) | 18 | 3
White blood cell count decreased (Investigations) | 7 | 15
White blood cell count increased (Investigations) | 21 | 6
White blood cells urine positive (Investigations) | 10 | 2
Decreased appetite (Metabolism and nutrition disorders) | 27 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 1
Dizziness (Nervous system disorders) | 4 | 5
Headache (Nervous system disorders) | 8 | 0
Insomnia (Psychiatric disorders) | 8 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 2
Rash (Skin and subcutaneous tissue disorders) | 33 | 3
Hypertension (Vascular disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT02545075/SAP_000.pdf
  • Study Protocol (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT02545075/Prot_001.pdf